CLINICAL TRIAL: NCT02020434
Title: A Phase 1, Open-label, Single-dose Study to Determine the Safety and Pharmacokinetics of Carbavance™ (RPX2014/RPX7009) in Subjects With Renal Insufficiency
Brief Title: The Safety and Pharmacokinetics of Carbavance™ (RPX2014/RPX7009) in Subjects With Renal Insufficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rempex Pharmaceuticals (a wholly owned subsidiary of The Medicines Company) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rempex 504
Record Dates: First submitted 2013-12-10; First posted 2013-12-25 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Subjects With Varying Degrees of Renal Insufficiency and; Subjects With Normal Renal Function
MeSH Terms: interventions — RPX7009

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single dose of RPX7009 and RPX2014 (Experimental): Single dose of combination RPX7009 and RPX2014
  Interventions: Drug: RPX7009 and RPX2014

INTERVENTIONS:
Drug: RPX7009 and RPX2014 — The study is designed to enroll approximately 32 subjects. There will be approximately 24 subjects with varying degrees of renal insufficiency and approximately 8 subjects with normal renal function.

SUMMARY:
RPX7009(beta-lactamase inhibitor) is being studied in combination with carbapenem (RPX2014)to treat bacterial infections, including those due to multi-drug resistant bacteria.

DETAILED DESCRIPTION:
The worldwide spread of resistance to antibiotics among Gram-negative bacteria, particularly members of the ESKAPE group of pathogens, has resulted in a crisis in the treatment of hospital acquired infections. In particular, the recent dissemination of a serine carbapenemase (e.g., KPC) in Enterobacteriaceae in US hospitals now poses a considerable threat to the carbapenems and other members of the beta-lactam class of antimicrobial agents.

Rempex is developing a fixed combination antibiotic of a carbapenem (RPX2014) plus a new beta-lactamase inhibitor (RPX7009) which has activity against serine beta-lactamases, including KPC. This Phase 1 study will assess the safety, tolerability and pharmacokinetics of intravenous RPX2014 and RPX7009, administered in combination in subjects with varying degrees of renal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18 through 80 years of age
2. Willing to abstain from alcohol for 48 hours prior to dosing through discharge
3. Normal volunteer first matched by age (± 10 years), BMI (± 20%), and gender to the mean values of the moderate renal insufficiency group.
4. Have negative test results for HBsAg, anti-HCV antibody and anti-HIV antibody.
5. Voluntarily consent to participate in the study
6. Sexually abstinent or agree to use two approved methods of contraception.
7. Assessment of renal insufficiency for assignment to study groups will be based on measurements of eGFR calculated by the MDRD equation at the Screening Visit to determine eligibility.

Exclusion Criteria:

1. Unstable or new medical conditions (e.g., cardiovascular, respiratory, hepatic, renal, gastrointestinal, autoimmune, endocrine, or neurological disorders)
2. Hypersensitivity or idiosyncratic reaction to β-lactam antibiotics (e.g. penicillins, cephalosporins, or carbapenems)
3. History of clinically significant seizures, head injury, or meningitis.
4. Current evidence or history of malignancy, excluding basal cell carcinoma, in the 2 years prior to Day -1 with no evidence of recurrence.
5. Females who are pregnant, lactating, or have a positive pregnancy test
6. Previously received any dose of Carbavance (RPX2014/RPX7009).
7. Current participation in another investigational study or participation in another investigational clinical study within 30 days prior to the Screening Visit.
8. Blood donation or significant blood loss (i.e., > 500 mL) within 56 days prior to Day 1.
9. Plasma or platelet donation within 14 days prior to Day -1.
10. Any acute illness requiring antibiotic drug therapy within 30 days prior to Day 1 or a febrile illness within 7 days prior to Day 1.
11. Vigorous exercise from 48 hours prior to Day -1 until the day of discharge from the study.
12. Positive urine drug/alcohol test at the Screening Visit or Day -1
13. Concurrent use of medications known to affect the elimination of serum creatinine (e.g., trimethoprim/sulfamethoxazole [Bactrim®] or cimetidine [Tagamet®]) and competitors of renal tubular secretion (e.g., probenecid) within 30 days prior to the first dose of study drug
14. Abnormal and clinically significant findings on physical examination, medical history, serum chemistry, hematology, or urinalysis
15. Use of any other prescription or nonprescription drugs, vitamins, grapefruit/grapefruit juice or dietary or herbal supplements within 14 days prior to Day -1.

    1. Oral contraceptives are permitted for birth control.
    2. Acetaminophen (≤ 1 g/day) and low-dose ASA (i.e., ≤ 325 mg per day) are permitted.
16. Currently receives hemodialysis or peritoneal dialysis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Safety from baseline through the end of the study | 7days
  Number of patients with adverse events; assessed by patient reporting, collection of vital signs, ECGs and absolute values and changes over time of hematology, chemistry and urinalysis

CONTACTS AND LOCATIONS:
Overall Officials: Chris Galloway, MD, Principal Investigator — Da Vita Clinical Research; Jolene K Berg, MD, Principal Investigator — Da Vita Clinical Research
Locations (2):
- United States (2):
  - DaVita Clinical Research, Lakewood, Colorado
  - DaVita Clinical Research, Minneapolis, Minnesota

REFERENCES:
- [Derived] Rubino CM, Bhavnani SM, Loutit JS, Lohse B, Dudley MN, Griffith DC. Single-Dose Pharmacokinetics and Safety of Meropenem-Vaborbactam in Subjects with Chronic Renal Impairment. Antimicrob Agents Chemother. 2018 Feb 23;62(3):e02103-17. doi: 10.1128/AAC.02103-17. Print 2018 Mar. PMID 29311069